CLINICAL TRIAL: NCT01483313
Title: Intelligence Performance in Adolescence After Early Exposure to Anesthesia and Minor Surgery
Brief Title: Intelligence Changes Following Minor Surgery
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled.
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, diansan su, Principal Investigator, RenJi Hospital
Other Study IDs: RenJiH-20111005
Record Dates: First submitted 2011-10-13; First posted 2011-12-01 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2012-03

CONDITIONS: Hypospadia; Phimosis; Inguinal Hernia
Keywords: Anesthestics; Minor surgery; Wechsler Intelligence Scale for Children; Cognitiion
MeSH Terms: conditions — Hypospadias; Phimosis; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Animal studies showed that many general anesthetics might result in neuron apoptosis and neurocognitive impairment in the developing brain. However results from human studies are conflicted. In present study, the investigators examined the association between early exposure to anesthesia and surgery for minor surgery and intelligence changes in adolescence using the Wechsler Intelligence Scale for Children.

ELIGIBILITY:
Inclusion Criteria:

1. Born from 1995
2. Male
3. Parents or guardian agree to attend this study
4. Undergone minor surgery (Repair of hypospadias, phimosiectomy, cryptorchidectomy or cryptorchidopexy and repair of inguinal hernia)
5. Children who scarify the No.1 to No.3 but no experience of any surgery.
6. Those who undergone minor surgery in Renji Hospital 4-6years ago.

Exclusion Criteria:

1. Any congenital central nervous system diseases
2. Any congenital heart diseases
3. Any congenital dysgnosia
4. Birth weight less than 2kg
5. Ever been hypoxic encephalopathy when birth

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators would like chose the Children who undergone minor surgery in Renji hospital 4-6years ago and their friends who never had any surgery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children | Average 5 years after surgery
  Wechsler Intelligence Scale for Children will be done after surgery, the expected average of 5 years after surgery.

SECONDARY OUTCOMES:
Achenbach Child Behavior Checklist | Average 5 years after surgery
  Wechsler Intelligence Scale for Children will be done after surgery, the expected average of 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, M.D., Ph.D, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China